CLINICAL TRIAL: NCT02085434
Title: Pediatric Practice-based Obesity Intervention to Support Families: FITLINE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Lori Pbert, Professor of Medicine, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H00000948
Record Dates: First submitted 2014-02-20; First posted 2014-03-12 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FITLINE practice-based referral program (Experimental)
  Interventions: Behavioral: FITLINE practice-based referral program
- Contemporaneous control (No Intervention)

INTERVENTIONS:
Behavioral: FITLINE practice-based referral program — The FITLINE practice-based referral program provides pediatric practices an easily accessible resource to help families make AAP-recommended Stage 1 lifestyle changes. The program includes a pediatric practice-based component (systems to identify overweight and obese children ages 8-12, a brief pediatric provider-delivered intervention, referral to the FITLINE counseling program, and feedback from the FITLINE nutritionist) and a parent support component(eight weekly FITLINE counseling telephone calls delivered by centrally located nutritionists). Providers receive a summary from the nutritionist of the progress made by families so they may support maintenance of an improved lifestyle, or refer for additional intervention.
  Arms: FITLINE practice-based referral program

SUMMARY:
The American Academy of Pediatrics (AAP) recommends a staged approach for pediatric practices to manage the growing problem of pediatric overweight and obesity, starting with Stage 1, Prevention Plus, which encourages families to improve basic lifestyle choices related to eating and activity in order to improve BMI status. This study will test the effectiveness of an innovative FITLINE telephone counseling program for overweight and obese 8-12 year olds seen in pediatric practices where nutritionists coach parents in improving their child's diet and physical activity, to reduce BMI. If found to be effective, the FITLINE program will provide a model for widespread implementation of Stage 1, Prevention Plus of the AAP expert committee recommendations through pediatric practices nationwide.

DETAILED DESCRIPTION:
The American Academy of Pediatrics (AAP) recommends a staged approach to the management of pediatric overweight and obesity, starting with Stage 1, Prevention Plus, which encourages families to improve lifestyle choices related to eating and activity in order to improve BMI status. Most pediatric practices, however, have difficulty implementing these guidelines due to limited time and access to weight loss experts to whom they can refer their patients and families, and burden to families in accessing in-person weight loss services. In response, The investigators team developed the FITLINE pediatric practice-based referral program that provides practices an easily accessible resource to help families make AAP-recommended Stage 1 lifestyle changes. The program includes two components. The first, a pediatric practice-based component, consists of systems to identify overweight and obese children ages 8-12, a brief pediatric provider-delivered intervention, referral to the FITLINE counseling program, and feedback from the FITLINE nutritionist. The second, a parent support component, consists of six weekly FITLINE counseling telephone calls delivered by centrally located nutritionists who provide tailored, personalized coaching, along with a parent booklet to guide parents in setting goals and working with their child to make Stage 1 lifestyle changes. Providers receive a summary from the nutritionist of the progress made by families so they may support maintenance of an improved lifestyle, or refer for additional intervention. A nonrandomized intervention study with contemporaneous control was used. Parents and their children ages 8-12 with BMI ≥85th percentile (N=40) were recruited from two pediatric practices. Practices implemented systems to identify overweight/obese children, prompt brief provider intervention, and refer parents to 6-weekly FITLINE telephone counseling sessions with a nutritionist who guided parents in setting goals and helping their child make American Academy of Pediatrics (AAP)-recommended lifestyle changes. Child BMI and parent survey of child diet and physical activity were completed at baseline and 3 months. Medical record data from 44 children matched for age and BMI was collected.

ELIGIBILITY:
Inclusion Criteria:

* child ages 8-12
* child BMI > 85th percentile for age/sex
* access to a telephone and parent available to participate in telephone counseling sessions,
* referred by the child's primary care provider (i.e., family deemed by the provider as able to participate in the study and interventions). If more than one child in a family is eligible, the oldest child will be invited to participate.

Exclusion Criteria:

* planning to move out of the area during the period of study participation
* medical condition that precludes adherence to AAP dietary and physical activity recommendations
* prescribed medications associated with weight gain, or (4) morbidly obese (> 300 pounds).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Baseline and 3 months post-baseline
  The child's weight and height were measure in the clinic using standard methodology. BMI was calculated from weight (kg)/height squared (in meters) and BMI-z score for age/sex determined using Centers for Disease Control growth charts.

SECONDARY OUTCOMES:
Diet | Baseline and 3-months post-baseline
  Parents completed a survey assessing: (1) parent's feeding style using an 11-item questionnaire to assess interactions of the parent with the child during the dinner meal; (2) parent's perceived support and barriers to addressing their child's behavior changes using the Caregiver Attitudes and Beliefs Survey, created by the authors; (3) a 12-item survey regarding number of days their child engaged in key dietary behaviors (e.g., eat breakfast in the morning, eat fast food or restaurant meal, eat dinner with the family, (4) number of days in past week their child ate 5 fruit or vegetables, and drank water, fruit juice, and punch/sweet tea/soda/sports drinks; and (5) type of milk the child drinks.
Physical activity behaviors | Baseline and 3 months post-baseline
  Parents completed a survey assessing: (1) parent's perceived support and barriers to addressing their child's behavior changes using the Caregiver Attitudes and Beliefs Survey, created by the authors; (2) a 12-item survey regarding number of days their child engaged in key physical activity behaviors (e.g., use computer or play video games, watch television, play sports).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States